CLINICAL TRIAL: NCT00079040
Title: A Phase II Study of Cisplatin Plus Etoposide (PE) Plus Bevacizumab (NSC #704865) for Previously Untreated Extensive Stage Small Cell Lung Cancer
Brief Title: Cisplatin, Etoposide, and Bevacizumab in Treating Patients With Previously Untreated Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02944; NCI-2012-02944 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E3501; E3501 (Other: Eastern Cooperative Oncology Group); E3501 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2012-12

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — Cisplatin; Etoposide; Bevacizumab

ARMS (1):
- Treatment (cisplatin, etoposide, bevacizumab) (Experimental): Chemotherapy: Patients receive cisplatin IV over 30-60 minutes on day 1 and etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Bevacizumab therapy: Beginning concurrently with chemotherapy, patients receive bevacizumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 17 courses (1 year) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: etoposide; Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving cisplatin and etoposide together with bevacizumab works in treating patients with previously untreated extensive-stage small cell lung cancer. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or deliver tumor-killing substances to them. Giving chemotherapy with a monoclonal antibody may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the combination of PE plus concurrent and sequential bevacizumab with respect to six month progression free survival in patients with previously untreated SCLC.

II. To evaluate the combination of PE plus concurrent and sequential bevacizumab with respect to survival and response rate.

III. To evaluate toxicity in patients with extensive small cell lung cancer, treated with the combination of PE plus concurrent and sequential bevacizumab who have received no prior systemic chemotherapy.

SECONDARY OBJECTIVES:

I. To determine if pre-treatment levels of plasma VEGF predict response to chemotherapy with Etoposide-Cisplatin plus concurrent + sequential bevacizumab.

II. To determine if pre-treatment plasma VEGF is predictive of progression free survival and overall survival in advanced SCLC.

III. To determine whether elevated plasma levels of endothelial cell-specific proteins (VCAM, E-selectin), reflective of chemotherapy or bevacizumab induced endothelial damage, are useful markers in assessing response to Etoposide/Cisplatin plus concurrent + sequential bevacizumab.

IV. To determine whether pre- and post-treatment plasma levels of basic fibroblast growth factor (bFGF) is predictive of progression free survival and overall survival or predictive of response to therapy.

OUTLINE: This is a multicenter study.

Chemotherapy: Patients receive cisplatin IV over 30-60 minutes on day 1 and etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Bevacizumab therapy: Beginning concurrently with chemotherapy, patients receive bevacizumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 17 courses (1 year) in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 weeks for up to 3 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histologic (or cytologic) proof of small cell lung cancer must be confirmed
* Patients must be clinically staged as extensive disease
* Patients must have measurable disease as defined by RECIST criteria; baseline scans/evaluation used to document measurable disease must be done within 4 weeks prior to registration; patients with measurable disease only or with both measurable and non-measurable disease are eligible
* Patients must have ECOG performance status of 0, 1, or 2
* Patients may not have had prior chemotherapy, immunotherapy, or biological therapy for lung cancer; previously irradiated lesions must not be the only site of measurable disease
* ANC > 1500/mm^3
* Platelets >= 100,000/mm^3
* Creatinine =< 1.5 mg
* Total bilirubin =< 1.5 mg
* Pregnant or breastfeeding women are excluded from the study because the agents used in this study may be teratogenic to a fetus or child and there is no information on the excretion of the agents or their metabolites into breast milk; all females of childbearing potential must have a blood test or urine study within 2 weeks, prior to registration to rule out pregnancy
* Women of childbearing potential and sexually active males are strongly advised to use an effective method of contraception
* Patients must be disease-free for > 5 years if they have a history of prior malignancies (except for cured basal or squamous cell skin cancers, or carcinoma in situ of the cervix)
* Patients must be considered on psychosocial grounds to be willing and able to comply with the requirements of treatment and follow-up
* Patients must not have CNS metastases; a head CT is required within 4 weeks prior to study entry for evaluation (MRIs are also acceptable)
* Urine dipstick for proteinuria of less than 1+ is required within 7 days prior to study entry; if urine dipstick is >= 1+ then a 24 hour urine for protein must demonstrate =< 1 gm of protein in 24 hours to allow participation in the study; NOTE: Urinalysis is also acceptable
* Patients must have INR =< 1.5 and a PTT no greater than the institutional upper limit of normal within 1 week prior to registration
* Patients must not have ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not have history of thrombotic or hemorrhagic disorders; patients must not have recently (within 6 months of registration) experienced arterial thromboembolic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, or myocardial infarction (MI); patients must also not have clinically significant peripheral artery disease
* Patients with history of hypertension must be well-controlled (=< 150/85) on a stable regimen of anti-hypertensive therapy
* Patients must not be receiving chronic daily treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory agents known to inhibit platelet function; treatment with dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and/or cilostazol (Pletal) is also not allowed
* Patients must not have serious non-healing wound, ulcer, or bone fracture, or major surgical procedure within 28 days prior to starting treatment; patients must not have had minor surgery or needle biopsies within 7 days of treatment
* Patients must not be on therapeutic anticoagulation
* Patients with a history of gross hemoptysis (defined as bright red blood of a 1/2 teaspoon or more) will be excluded from this trial
* Patients must have had no prior radiation therapy to the site of evaluable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Sandler, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between June 8, 2004 and August 18, 2006.
Groups:
- Cisplatin, Etoposide, Bevacizumab: Cisplatin 60 mg/m2 IV, Etoposide 120 mg/m2 IV, and Bevacizumab 15 mg/kg IV on Day 1, Etoposide 120 mg/m2 IV on days 2 and 3 of a 21-day cycle for 4 cycles. Bevacizumab continued for 1 year or until progression.
Period: Overall Study
Arm/Group | Cisplatin, Etoposide, Bevacizumab
Started | 65
Completed | 63
Not Completed | 2
Not completed — Withdrew before treatment | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin, Etoposide, Bevacizumab
Number analyzed (Participants) | 63
Age, Continuous [Median (Full Range); unit: Years] | 65 [45 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive and Progression-free (PF) at 6 Months
Description: Progression-free survival was defined to be the interval in months from the date of registration to the date of documented disease progression or to death without progression. Patients alive without progression at 6 months were included in the numerator when calculating the progression-free rate.
Time Frame: 6 months
Population: Per protocol, the analysis included all eligible, treated patients (n=63). The safety analysis included all treated patients, regardless of eligibility (n=64).
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cisplatin, Etoposide, Bevacizumab
Number analyzed (Participants) | 63
Percentage of Participants | 30.2 [19.3 to 43.1]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from registration to death or date last known alive. Patients alive at last follow-up are censored.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 1 year
Population: Per protocol, the analysis included all eligible, treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin, Etoposide, Bevacizumab
Number analyzed (Participants) | 63
months | 10.9 [7.9 to 12.2]

3. Secondary Outcome: Best Objective Response
Description: Number of patients with complete or partial response by RECIST criteria.
Time Frame: Assessed every 6 weeks
Population: Per protocol, the analysis included all eligible, treated patients.
Measure: Number; unit: Patients Responding
Arm/Group | Cisplatin, Etoposide, Bevacizumab
Number analyzed (Participants) | 63
Patients Responding | 40 [50.4 to 75.6]
Statistical Analysis 1: Comparison: Cisplatin, Etoposide, Bevacizumab; Test type: Superiority or Other; Percentage = 63.5, 90% CI 2-sided [52.4 to 73.6]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at each treatment visit (approximately every 3 weeks) and through 30 days following the end of treatment
Description: Assessment was done routinely for the safety population, which consisted of all 64 treated patients.
Arm/Group | Cisplatin, Etoposide, Bevacizumab
Serious Adverse Events (participants affected / at risk) | 49/64
Other Adverse Events (participants affected / at risk) | 63/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin, Etoposide, Bevacizumab (N=64)
Allergic Reaction (Immune system disorders) | 1
Low Hemoglobin (Blood and lymphatic system disorders) | 3
Low Leukocytes (Blood and lymphatic system disorders) | 19
Lymphopenia (Blood and lymphatic system disorders) | 1
Low Neutrophils (Blood and lymphatic system disorders) | 37
Low Platelets (Blood and lymphatic system disorders) | 9
Sinus Bradycardia (Cardiac disorders) | 1
Cardiac ischemia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 5
Hypotension (Cardiac disorders) | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 1
Cardiac - other (Cardiac disorders) | 1
Fatigue (General disorders) | 8
Death - multiorgan failure (General disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1
Muco/stomatitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdomen, hemorrhage (Gastrointestinal disorders) | 1
Bronchopulmonary, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Febrile Neutropenia (Infections and infestations) | 3
Infection w/ gr 3-4 neutrophils, lung (Infections and infestations) | 1
Infection w/ gr 0-2 neutrophils, lung (Infections and infestations) | 1
Infection w/ gr 3-4 neutrophils, blood (Infections and infestations) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 7
Extremity, lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic generalized weakness (General disorders) | 1
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 1
Bone, pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 3
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1
Pain, other (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/upper respiratory, other (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin, Etoposide, Bevacizumab (N=64)
Hemoglobin (Blood and lymphatic system disorders) | 4
Leukocytes (Blood and lymphatic system disorders) | 40
Neutrophils (Blood and lymphatic system disorders) | 33
Platelets (Blood and lymphatic system disorders) | 28
Hypertension (Cardiac disorders) | 9
Hypotension (Cardiac disorders) | 7
Fever w/o neutropenia (Infections and infestations) | 7
Insomnia (General disorders) | 6
Rigors/chills (General disorders) | 7
Weight loss (General disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 47
Injection site reaction (Skin and subcutaneous tissue disorders) | 4
Pruritis/itching (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Anorexia (Gastrointestinal disorders) | 28
Constipation (Gastrointestinal disorders) | 30
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 17
Dysphagia (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 10
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 14
Muco/stomatitis (symptom), oral cavity (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 43
Taste disturbance (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 18
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 6
Alkaline phosphatase (Metabolism and nutrition disorders) | 12
AST, SGOT (Metabolism and nutrition disorders) | 13
Hypercalcemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 9
Creatinine (Metabolism and nutrition disorders) | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 21
Hyperkalemia (Metabolism and nutrition disorders) | 10
Hypokalemia (Metabolism and nutrition disorders) | 11
Proteinuria (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 26
Dizziness (Nervous system disorders) | 6
Neuropathy, motor (Nervous system disorders) | 5
Neuropathy, sensory (Nervous system disorders) | 17
Vision - blurred (Eye disorders) | 5
Back, pain (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 10
Muscle, pain (Musculoskeletal and connective tissue disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less